CLINICAL TRIAL: NCT03072745
Title: Distinct Effect of Insomnia on Cognitive Performance in Individuals With Complex Chronic Pain
Brief Title: Insomnia and Cognitive Performance in Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2010/182
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Chronic Pain; Insomnia
Keywords: Cognitive Impairment
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuropsychological assessment (Experimental): Assessment with a neuropsychological test battery and self-report measures.
  Interventions: Diagnostic Test: Neuropsychological assessment

INTERVENTIONS:
Diagnostic Test: Neuropsychological assessment — Assessment with a neuropsychological test battery examining different aspects of memory and executive functioning

SUMMARY:
The aim of the present study is to examine cognitive function in a patient population with complex chronic pain to test the hypothesis that insomnia severity on its own predicts objective cognitive function, and that a correlation is not better explained by comorbid depression or anxiety, morphine equivalent daily dose, or the level of pain itself.

DETAILED DESCRIPTION:
Almost 20 % of the adult European population suffers from chronic pain of moderate to severe intensity, and clinical insomnia has been reported in 53-73% of chronic pain patients. Insomnia seems to be correlated with small to moderate impairments in several cognitive functions involved in working and episodic memory and in attention tasks, and chronic pain has been shown to be associated with objective deficits in memory and executive functioning. The aim of the present study is to examine cognitive function in a patient population with complex chronic pain to test the hypothesis that insomnia severity on its own predicts objective cognitive function, and that a correlation is not better explained by comorbid depression or anxiety, morphine equivalent daily dose, or the level of pain itself.

Inividuals with complex chronic pain are assessed with a neuropsychological test battery examining different aspects of memory and executive functioning:

The Digit Span subtest from Wechsler's Adult Intelligence Scale III (WAIS-III): Verbal working memory.

Claeson-Dahl Inventory of Learning and Memory (CD): Verbal retention. The Rey Complex Figure Test (RCFT): Visuospatial retention. The Wisconsin Card Sorting Test (WCST): Cognitive flexibility. The Trail-Making Test (TMT): Sustained attention.

The presence of insomnia is examined with the Bergen Insomnia Scale (BIS) , and insomnia severity with the Insomnia Severity Index (ISI). Present pain level at the time of the neuropsychological assessment is quantified using the Visual Analogue Scale (VAS). Pain medication is transformed to the morphine equivalent daily dose (MEDD). Anxiety and depression are assessed with the Hospital Anxiety and Depression Scale.

ELIGIBILITY:
Inclusion Criteria:

* Attending tertiary chronic pain management

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-05-01 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Memory impairment | 1 day
  Composite score comprising verbal working memory, verbal retention, and visuospatial retention.

SECONDARY OUTCOMES:
Executive functioning impairment | 1 day
  Composite score comprising cognitive flexibility and sustained attention.

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Gordh, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided